CLINICAL TRIAL: NCT05431439
Title: Omics of Cancer: OncoGenomics
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000046; 000046-C
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms; Cancer
Keywords: Oncogenomics; Malignancies; Therapeutic Strategies; Human Genome Project; Cancer; Tumor Genome; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with cancer or cancer predisposition

SUMMARY:
Background:

Cancer is a leading cause of death in the United States. Researchers want to know more about how cancer develops and grows. They want to understand more about cancers that run in families. This information will help them find better ways to diagnose and treat cancer. Researchers need to collect data from many people who either have cancer or who may get cancer.

Objective:

To establish a registry of data about people with cancer. The natural history registry will be linked to a database with information about their genetics.

Eligibility:

People aged 4 weeks and older with a diagnosis of any cancer. People with precancerous conditions or with a family history of an inherited cancer are also needed.

Design:

Participants will answer questions about their medical history. This visit can be in-person or by phone.

Participants will provide blood and saliva samples. Researchers will also collect any samples the participants may already have given in the past. These may include tumor biopsies or samples of bone marrow or other body fluids. No blood will be collected from children younger than 3 years.

No new surgeries or biopsies will be done for this study.

The samples will be used for genetic research.

Researchers will follow up with participants once a year. They will get an updated medical history. They will ask for any new biopsies or other tissue samples. They may collect new saliva and blood samples.

Participants may continue in the study for the rest of their lives....

DETAILED DESCRIPTION:
Background

* Cancer is the second leading cause of disease-related mortality in the US and the primary leading cause of US disease-related mortality in individuals aged 40-79
* One of the missions of the Oncogenomics Section is to identify new targets and develop new therapeutic strategies for currently incurable malignancies as well as to improve the quality of life for adults and children with cancer. Overall, approximately 1,918,030 individuals, 983,160 males, and 934,870 females will be diagnosed with cancer in 2022

Objective

-To establish a registry in which clinical data of participants with cancer or cancer predisposition is linked to the genomic database of analyzed samples

Eligibility

* Age >= 4 weeks
* Participants must have a diagnosis of any tumor, malignancy, pre-malignant disorder, or evidence of an inherited cancer syndrome based on family history and/or other manifestations of the syndrome (i.e., polyposis, plexiform neurofibromas, myelodysplastic syndrome
* Participants must have biospecimen (e.g., including tumor, normal, blood, bone marrow, serum, plasma, or any other specimen) that has been previously collected and is available for research analysis, be scheduled to undergo surgery or biopsy for routine patient care on another research or standard of care protocol or be willing to provide blood and/or saliva specimens. Note: blood will not be drawn in children < 3 years old

Design

* Participants will be enrolled at NIH
* Collected samples will be studied to:

  * Examine tumor samples for oncogenic drivers using next-generation whole genome sequencing (WGS), whole exome sequencing (WES), panel, or RNA sequencing
  * Analyze germline samples for known or novel cancer predisposition genes using WGS, WES, or panel sequencing
  * Determine the feasibility of longitudinal collection and analyses of liquid biopsies alongside the analysis of matched tumor samples
  * Establishment of Epstein-Barr virus (EBV) transformed cell lines from blood and/or bone marrow for medical research
  * New methodologies such as proteomics and metabolomics analysis in the investigation of cellular, molecular, genetic, and genomic biology, to probe for new therapeutic targets, and to develop new treatment approaches
* Expected accrual 50-500 participants per year. Total protocol accrual goal 5,000 participants

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 4 weeks
* Participants must have:

  * diagnosis of any tumor, malignancy, pre-malignant disorder

OR

* evidence of an inherited cancer syndrome based on family history and/or other manifestations of the syndrome (i.e., polyposis, plexiform neurofibromas, myelodysplastic syndrome)

  -Participants must
* have biospecimen (e.g., tumor, normal, blood, bone marrow, serum, plasma, or any other specimen) that has been previously collected and is available for research analysis

OR

--be scheduled to undergo surgery or biopsy for routine patient care on another research or standard of care protocol

OR

--be willing to provide blood and/or saliva specimens. Note: does not apply to children < 3 years old

-The ability of participant or parent/guardian to understand and the willingness to sign a written consent document.

EXCLUSION CRITERIA:

None

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a trial to establish a registry in which clinical data of participants with cancer or cancer predisposition is linked to a database of analyzed samples. Participants will be enrolled in the protocol at the NIH Clinical Center from the NIH CC patient population or or from referrals from an extramural facility or treating physicians.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
establish a registry in which clinical data of participants with cancer or cancer predisposition is linked to the genomic database of analyzed samples | 20 yrs
  perform systematic genetic and genomic analysis to enrolled participants treated at the Center for Cancer Research (CCR, NCI) and all Divisions of NCI for the identification of biomarkers and targets of potential therapeutic actionability

SECONDARY OUTCOMES:
determine the feasibility of longitudinal collection and analyses of liquid biopsies alongside the analysis of matched tumor samples | Ongoing throughout study
  to characterize heterogeneity and to identify therapeutically resistant clones
examine tumor samples | Ongoing throughout study
  oncogenic drivers using next-generation whole genome (WGS), exome (WES), and/or RNA sequencing
analyze germline samples | Ongoing throughout study
  known or novel cancer predisposition genes using WGS, WES, and/or RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Javed Khan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@ In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000046-C.html